CLINICAL TRIAL: NCT04664543
Title: Efficacy of Free Versus Low Residue Diet as Preparation for Screening Colonoscopy: CriLi Study, a Pilot Trial
Brief Title: Efficacy of Free Versus Low Residue Diet as Preparation for Screening Colonoscopy
Acronym: CriLi
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organization and logistic problems due to COVID19 pandemy
Sponsor: Parc Taulí Hospital Universitari (Other)
Collaborators: Consorci Sanitari de Terrassa (Other); Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, Salvador Machlab, Principal Investigator, Parc Taulí Hospital Universitari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2019307
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer; Colon Polyp; Colon Adenoma
Keywords: colonoscopy; bowel cleansing; low fiber diet; colonoscopy preparation
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 days of low residue diet (Active Comparator): Currently participants in the colorectal cancer screening program follow a 3 days low residue diet before colonoscopy. This is the active comparator arm of this study.
  Interventions: Other: Three days low residue diet
- Free diet (Experimental): Participants assigned to this arm are NOT instructed to follow any kind of restriction in the diet before colonoscopy.
  Interventions: Other: Free diet

INTERVENTIONS:
Other: Free diet — To follow the regular dietary habits with no restriction nor modification.
  Other Names: Liberal diet, habitual diet
  Arms: Free diet
Other: Three days low residue diet — To follow the three days before colonoscopy a diet with low content in fiber or residues.
  Other Names: low fiber diet
  Arms: 3 days of low residue diet

SUMMARY:
One tricky aspect of the recommendations for colonoscopy prep is diet. This has a significant impact on the experience of the patient or participant in the screening program and, on the other hand, low adherence has been found in some studies despite a potential Hawthorne effect . It is noteworthy that despite its impact on patient experience, it is an area for which little evidence is available, which is why the guidelines give low-quality recommendations and there is probably considerable variability in clinical practice .

In the early days of colonoscopy, a liquid diet for 48 hours was mainly recommended, although some centers indicated a low-residue diet or even the commercially available NASA astronaut diet. Later, the indication for a liquid diet was consolidated until finally numerous studies were published in favor of a low-residue diet, managing to increase tolerance and the quality of the preparation . A limitation of the preparation studies must be borne in mind that the colon cleansing rating scales were not introduced until 1999 when the Aronchick scale was published.

Although there is solid evidence in favor of a low-residue diet versus a liquid diet, the investigators do not have evidence on how many days of a low-residue diet should be recommended, and this is reflected in the ESGE (European Society of Gastrointestinal Endoscopy) and ASGE (American Society of Gastrointestinal Endoscopy) guidelines . A randomized clinical trial comparing 3 days versus 1 day of a low residue diet has recently been published . There were no statistically significant differences in the rate of adequate preparations (82.7% vs. 85.6% OR 1.2 95% IC 0.72 to 2.15). However, this study has limited statistical power and a design that allows a non-inferiority analysis has not been followed. In relation to this, our research group is finalizing a non-inferiority clinical trial in whose intermediate analysis, with 421 participants, the non-inferiority of 1 day of diet is fulfilled (rate of poor preparation in 1 day 0.95% vs. 4.74% in 3 days; d + 5%, difference -3.78% IC -6.88% to -1.12%) (38).

It is likely, taking into account the available evidence and its evolution, that diet plays a secondary role in preparation. Although no studies designed to directly assess this have been conducted, the research group has indirect data.

Walter et al, under the hypothesis that the impact of the fractional preparation and the new preparations on the preparation diminished the importance of the diet, conducted a non-inferiority clinical trial between 2012 and 2013 in which they randomized the patients to follow a diet liquid versus low residue for one day and fractional preparation with Moviprep (39). They established a non-inferiority margin of -13.5%. Their results show a rate of good preparation (Boston> 5) in 68/72 (94.4%) in a liquid diet compared to 60/68 (88.2%) in a low-residue diet (p = 0.04) with a difference of -5.08% demonstrating non-inferiority of the low residue diet.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 50 and 69 years old.
* Participants in the Program for the Early Detection of Colorectal Cancer with a positive result in the test for detecting occult blood in feces
* That they accept a colonoscopy and that they agree to participate in the study.

Exclusion Criteria:

* Contraindication to performing a colonoscopy.
* Severe renal insufficiency (<30 ml / min).
* Known hypersensitivity or allergy to polyethylene glycol, ascorbic acid or sulfate.
* Known glucose-6-phosphate dehydrogenase deficiency.
* Known phenylketonuria.
* Known dyselectrolytemia: hyper / hyponatremia, hyperphosphatemia, hypermagnesemia, hyper / hypokalemia, hypocalcemia.
* Gastric emptying disorders: Known gastroparesis.
* Known hypoalbuminemia less than 3.4 g / dl.
* Crohn's disease or known ulcerative colitis.
* Participants with difficult-to-control hypertension (SBP> 170mmHg or TAD> 100mmHg) or NYHA grade III or IV heart failure.
* Ascites of any etiology
* People with cognitive impairment or mental illness that makes it difficult to adhere to instructions.
* People who do not understand Catalan or Spanish.
* Factors of poor preparation: liver cirrhosis, diabetes mellitus, treatment with tricyclic antidepressants, opioids or neuroleptics, limited mobility, chronic constipation, history of colon or intestinal resection (appendectomy is not an exclusion criterion), poor preparation in previous colonoscopy Parkinson's disease, multiple sclerosis.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Adequate bowel cleansing | During colonoscopy (At the withdrawal phase)
  Bowel cleansing has a rating using the Boston Bowel Preparation Scale above 1 in each segment . This score ranges fron 0 to 3 in each one of the three segments. Zero is the worst outcome and 3 is the best cleansing

SECONDARY OUTCOMES:
Diet tolerability | The day of the colonoscopy just before beginning
  Tolerance to the diet assigned to the participant measured with a likert scale from 0 to 5, 0 the worst ad 5 the best.
Preparation tolerability | The day of the colonoscopy just before beginning
  Tolerance to the cleansing solution used for bowel cleansing measured with a likert scale from 0 to 5, 0 the worst ad 5 the best.
Adenoma detection | adenoma detection is done during the colonoscopy but assesment will be done at the end of the study with the histology reports
  An adenoma was detected, resected and confirmed by the histology report in the colonoscopy.
Polyp detection | During colonoscopy
  Polyp detection in the colonoscopy as reported by the endoscopist.
Ceacal intubation time | During colonoscopy
  Time expended in reaching the cecum
Withdrawal time | During colonoscopy
  Time expended in the withdrawal from cecum till the anus.
Excellent cleansing | During colonoscopy
  Colonoscopy achieving a Boston Bowel Preparation Scale (BBPS) of at least 8 points or above. BBPS global score ranges from 0 to 9, being 9 the best cleansing outcome.
Information perceived quality | The day of the colonoscopy just before beginning
  Perceived quality of the instructions and education received for the colonoscopy. preparation by the participant. Assessed using a likert scale from 0 to 5. Five is the best outcome and 0 the worst.
Preparation quality in each segment | During colonoopy
  Boston Bowel Preparation Score in each segment, it ranges from 0 to 3 being 3 the best cleansing outcome and 0 the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Martínez, PhD, Study Director — Hospital Universitari Parc Taulí
Locations (1):
- Hospital Universitari Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Machlab Mashlab S, Martinez-Bauer E, Lopez P, Pujals MDM, Fernandez-Banares F, Selva A, Calvet X, Campo R. Unrestricted vs three-day low-residue diet for colonoscopy preparation. Results of a feasibility randomized trial. Rev Esp Enferm Dig. 2025 Jun;117(6):349-350. doi: 10.17235/reed.2024.10417/2024. PMID 38591600